CLINICAL TRIAL: NCT07277647
Title: The Effect of Head and Neck Stretching Exercises on Voice, Anxiety and Psychological Resilience After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, yasemin ay karadaş, PHD, Ataturk University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: B.30.2.ATA.0.01.00/359
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Effects of Post-Thyroidectomy Head and Neck Stretching Exercises on Voice, Anxiety, and Psychological Resilience
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is a quasi-experimental research with a pre-test-post-test control group. This research was conducted at the General Surgery Clinic of Atatürk University Research Hospital between May 2023 and January 2024. The population of this study consisted of patients who underwent thyroidectomy at the General Surgery Clinic of Atatürk University Research Hospital. The study sample consisted of all patients who were informed, agreed to participate, and met the inclusion criteria. The study was completed with 103 patients (training: 50, control: 53) who met the study criteria. The Patient Identification Form, Voice Handicap Index, State-Trait Anxiety Inventory, and Connor-Davidson Resilience Scale were used to collect the research data.Data Collection Process Patients undergoing thyroidectomy who agreed to participate in the study and met the sample selection criteria were included in the study. Patients undergoing thyroidectomy are generally admitted to the hospital one day before surg
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental): Structured patient education + neck stretching exercises
  Interventions: Behavioral: Structured patient education + neck stretching exercises
- Control Group (No Intervention): routine care only

INTERVENTIONS:
Behavioral: Structured patient education + neck stretching exercises — The intervention is a nurse-led, structured patient education program based on the, combined with a supervised head-neck stretching exercise program. Unlike routine postoperative care, this intervention includes: (1) preoperative individualized education using the Teach-Back method, (2) a printed educational booklet specifically developed for thyroidectomy patients, and (3) a standardized 30-day head-neck stretching exercise program initiated in the early postoperative period (starting on postoperative day 1). The exercise program is performed daily at home with visual and written guidance. In addition, patients receive regular follow-up and reinforcement during the postoperative period. This comprehensive and multimodal structure distinguishes the intervention from standard care and other single-component educational approaches.
  Arms: Education Group

SUMMARY:
The aim of this clinical randomized controlled trial is to evaluate the effects of head and neck stretching exercises performed after thyroidectomy on voice function, anxiety, and psychological resilience, and to examine the effectiveness of this intervention in adult patients undergoing thyroidectomy.

The primary questions to be answered are:

Do head and neck stretching exercises improve voice function (Voice Handicap Index) after thyroidectomy? Do head and neck stretching exercises reduce patients' anxiety levels and increase psychological resilience? As a comparison group, researchers will compare the effects of head and neck stretching exercises to a control group receiving only routine care to assess the effects of exercises on voice, anxiety, and psychological resilience.

Participants will be asked to participate in the following procedures:

Patients in the experimental group will undergo head and neck stretching exercises in the early post-thyroidectomy period.

Voice function, anxiety, and psychological resilience will be measured in both groups before surgery and at postoperative day 1, week 1, week 2, and month 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65, with adequate cognitive functions, who could communicate in Turkish, and who volunteered to participate in the study were included in our study.

Exclusion Criteria:

* Individuals who had previously undergone partial thyroidectomy, had cervical problems before thyroidectomy, had current or previous voice disorders, or had any illness that could affect decision-making ability (psychological disorder, dementia, etc.) were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
State Anxiety Level | Preoperative, postoperative 1st day, 1st week, 2nd week and 1st month.
  State anxiety level will be measured using the State-Trait Anxiety Inventory (STAI).

CONTACTS AND LOCATIONS:
Overall Officials: NEZİHA KARABULUT, Principal Investigator, Study Director — Ataturk University Faculty of Nursing, Erzurum, Türkiye
Locations (1):
- Atatürk University Research Hospital, Erzurum, Türkiye, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared in order to protect participant confidentiality and because the ethical approval for this study limits data use to the current research purposes only.